CLINICAL TRIAL: NCT05229978
Title: Engagement 2.0 Forms of Consent for Data (re-)Use
Acronym: ENGAGE
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: Engage 2.0
Record Dates: First submitted 2022-01-07; First posted 2022-02-08 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-05

CONDITIONS: Alzheimer Disease, Early Onset; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with AD or mild cognitive impairment due to AD: All three 'arms' take part in a focus group or interview. The conversation topics will be the same (with the aim to gauge interpretations / needs / thoughts / feelings with regard data usage for research and the role health data engagement interfaces (Dynamic Consent) may play in this.
  Interventions: Other: Showing an existing Dynamic Consent (computer interface) as prompt
- Informal carers of patients with AD or mild cognitive impairment due to AD: All three 'arms' take part in a focus group or interview. The conversation topics will be the same (with the aim to gauge interpretations / needs / thoughts / feelings with regard data usage for research and the role health data engagement interfaces (Dynamic Consent) may play in this.
  Interventions: Other: Showing an existing Dynamic Consent (computer interface) as prompt
- Dementia experts/specialists: Given their expertise on dementia from a professional point of view, a focus group is conducted with dementia specialists in order to elicit their views and ideas on health data engagement interface like Dynamic Consent.
  Interventions: Other: Showing an existing Dynamic Consent (computer interface) as prompt

INTERVENTIONS:
Other: Showing an existing Dynamic Consent (computer interface) as prompt — An existing Dynamic Consent interface will be shown as a prompt halfway through the focus group sessions.

SUMMARY:
The objective of this qualitative study is to create a better understanding of patients' mental model of health data engagement interfaces and tools (such as Dynamic Consent). The researchers will focus especially on those people who - plausibly - require adjusted communication particularities and interaction modalities due to a cognitive impairment stemming from a neurodegenerative disease. Taking into account the specific characteristics of patients with dementia, the goal of this study is to investigate how to communicate according to patients' personal skills and capabilities and identify both the proper support mechanisms for engagement 2.0 consent as well as feedback mechanisms (return of research results). Through a focus group & interview setup, this study will discern design requirements and propose design recommendations for the (future) development of health data engagement interfaces.

DETAILED DESCRIPTION:
While unprecedented amounts of multimodal health data become increasingly available and their secondary use in clinical and (bio)medical research holds great promise, people's agency over this data is in contention. In the context of biobank research, patient-centered initiatives such as 'dynamic consent' have been proposed as a way to provide people with ownership over their health data by allowing for granular expression of their consent preferences using a digital interface. Although such interfaces have been positively assessed within their original biobank context, more heterogeneous audiences will need to be considered if such a socio-technical tool is to be adopted widely and provide people ownership over their electronic medical records. One subset of people that will require adjusted functionalities and interaction modalities in this regard are those with a cognitive impairing condition like dementia, given the illness' consequences on decision making capacity. This study qualitatively explores the user & social requirements of a tool like dynamic consent if it is to be used in a meaningful way also by people with dementia and their (informal) carers. We report findings from interviews and an expert focus group with people with dementia, their caretakers, and experts to depict their views and requirements on a tool like dynamic consent.

ELIGIBILITY:
Inclusion Criteria:

* no diagnosed cognitive impairment but first-degree relative with AD
* mild cognitive impairment due to AD (diagnosed according to the NIA/AA diagnostic criteria)
* mild dementia due to AD (diagnosed according to the NIA/AA diagnostic criteria)

Exclusion Criteria:

* Patients with moderate to severe dementia due to AD, defined as MMSE total score 20/30 or lower

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients with mild MCI due to AD
  * Patient's with mild dementia due to AD
  * Subjects with no diagnosed cognitive impairment but first-degree relative with AD
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Qualitative data: interpretations / opinions / needs / thoughts / feelings with regard to clinical data usage and dynamic consent. | 1-2 months. During the focus groups and interviews, answers given by participants will be audiorecorded and later transcribed to be thematically analysed.
  Collected in response to questions from an open-ended questionnaire (interview guide), the outcome of the focus groups and interviews will be rich qualitative data that will provide a better understanding of patients' assumed skills, capabilities and preferences necessary to meaningfully interact with health data engagement (dynamic consent) interfaces" for clinical data usage consent.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Van den Bogaert, Master's, Principal Investigator — VUB (Vrije Universiteit Brussel)
Locations (1):
- Universitair Ziekenhuis Brussel (UZB), Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No
The qualitative data in this study (i.e. audio recordings from the focus groups and interviews) will be collected, stored and analysed only by the PI and the central contact backup.